CLINICAL TRIAL: NCT00959166
Title: A Prospective Case-control Study to Assess Neuroinflammation and Neurocognitive Function in Patients With Acute Hepatitis C and Chronic HIV Co-infection - a PET Study
Brief Title: To Assess Neuroinflammation and Neurocognitive Function in Patients With Acute Hepatitis C and Chronic HIV Co-Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09/H0712/17
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Acute Hepatitis C; HIV; HIV Infections
Keywords: Acute hepatitis C; HIV; Neurocognitive function; Neuroinflammation
MeSH Terms: conditions — HIV Infections; Neuroinflammatory Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV/acute HCV coinfection (Other): Subjects with HIV/acute HCV coinfection (aHCV cases) were required to have acute HCV, defined by a new positive plasma HCV RNA test within 12 months of a negative HCV RNA test.
  Interventions: Other: PET scan
- HIV mono (Other): HIV-infected individuals without hepatitis C co-infection
  Interventions: Other: PET scan

INTERVENTIONS:
Other: PET scan — PET brain scan

SUMMARY:
This study plans to evaluate what happens to the brain in patients with HIV and early hepatitis C. The investigators will be comparing 3 groups of individuals:

* Group 1: Individuals with HIV infection and acute (early) hepatitis C infection
* Group 2: Individuals with HIV infection
* Group 3: Healthy volunteers

DETAILED DESCRIPTION:
Subtle changes to the brain, which doctors find difficult to detect through conversation or examination, may occur in patients with HIV and/or hepatitis C infection. It is not currently known whether the brain is affected in early (or acute) hepatitis C.

Individuals wishing to take part will complete a series of tests assessing different aspects of their brain including:

* 2 brain scans using different technology:

  * Magnetic resonance imaging (MRI) brain scan with spectroscopy
  * CT PET brain scan
* A computer game test which measures brain function
* 2 short questionnaires

Results of these tests will be analyzed and compared between 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 antibody positive for at least 12 months
2. Acute HCV (Blood HCV PCR positive with negative PCR within past 8 months)
3. HCV genotype 1
4. Ability to give informed consent
5. Aged > 25 years
6. Male
7. Abbreviated Mental Test Score of at least 8/10

Exclusion Criteria:

1. Evidence of established cirrhosis or encephalopathy
2. Commencing or any change to HIV medications within 12 weeks
3. Active opportunistic infection
4. Taking anti-depressants or any psychoactive medications within past 4 weeks
5. Use of benzodiazepines within past 4 weeks
6. Recent significant head injury
7. Established dementia
8. Alcohol dependence or recreational drug misuse
9. Untreated early syphilis
10. Hepatitis B infection (HBsAg positive)
11. Pregnancy
12. Unable to give informed consent
13. Any contraindication to MR scanning

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garvey LJ, Pavese N, Ramlackhansingh A, Thomson E, Allsop JM, Politis M, Kulasegaram R, Main J, Brooks DJ, Taylor-Robinson SD, Winston A. Acute HCV/HIV coinfection is associated with cognitive dysfunction and cerebral metabolite disturbance, but not increased microglial cell activation. PLoS One. 2012;7(7):e38980. doi: 10.1371/journal.pone.0038980. Epub 2012 Jul 12. PMID 22808022

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV/Acute HCV Coinfection: Subjects with HIV/acute HCV coinfection
Period: Overall Study
Arm/Group | HIV/Acute HCV Coinfection | HIV Mono
Started | 24 | 57
Completed | 24 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV/Acute HCV Coinfection | HIV Mono | Total
Number analyzed (Participants) | 24 | 57 | 81
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [36 to 44] | 47 [39 to 56] | 44 [36 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 24 | 50 | 74
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 57 | 81
Time-elapsed since HIV diagnosis [Median (Inter-Quartile Range); unit: years] | 6 [3 to 12] | 11 [5 to 16] | 8.5 [3 to 16]
Current CD4+ cells [Median (Inter-Quartile Range); unit: cells/uL] | 590 [458 to 745] | 505 [382 to 783] | 547 [382 to 783]
Number of participants receiving antiretroviral therapy [Count of Participants; unit: Participants] | 17 | 54 | 71
Plasma HIV viral load below 50c/ml [Count of Participants; unit: Participants] | 16 | 54 | 70

OUTCOME MEASURES:

1. Primary Outcome: Association of 11C-labelled PK11195 Uptake Using PET With Acute HCV and HIV Infection
Description: Association of 11C-labelled PK11195 uptake using PET with acute HCV and HIV infection by PK11195 PET ligand binding. The ligand PK11195 is selective for the peripheral benzodiazepine binding site and exhibits minimal binding in normal brain. In brain lesions, however, there is a massive increase in binding.
Time Frame: 30 days
Population: 16 subjects in total had PET scans and were included in the PET outcome
Measure: Mean (Standard Deviation); unit: binding potential ratio
Arm/Group | HIV/Acute HCV Coinfection | HIV Mono
Number analyzed (Participants) | 8 | 8
binding potential ratio | 0.18 (0.10) | 0.22 (0.13)

2. Secondary Outcome: Ratio of NAA/Cr (N-acetyl Aspartate/Creatine) Cerebral Metabolites
Description: Association between patient characteristics and 11C-labelled PK11195 uptake using PET, CNS metabolite ratios.
  By quantifying the surrogate markers of N-acetylaspartate (NAA), creatine (Cr) offers insight into the neuronal integrity, cell membrane synthesis and turnover, macrophage infiltration, inflammation status, and levels of microglial activation and gliosis within the sampled CNS tissue.
Time Frame: 30 days
Population: 24/12 subjects in each study group had MR spectroscopy and could be included in this analysis
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HIV/Acute HCV Coinfection | HIV Mono
Number analyzed (Participants) | 24 | 12
ratio | 1.42 (0.25) | 1.35 (0.10)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | HIV/Acute HCV Coinfection | HIV Mono
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/57
Other Adverse Events (participants affected / at risk) | 0/24 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes